CLINICAL TRIAL: NCT00614471
Title: A Randomized, Open Label Study of the Effect of Peginterferon Alfa-2a (40KD) (PEGASYS®) Plus Entecavir (Baraclude®) Combination Therapy on Quantitative Changes in HBeAg in Treatment-naive Patients With HBeAg Positive Chronic Hepatitis B
Brief Title: A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) Plus Entecavir in Treatment-Naive Patients With HBeAg-Positive Chronic Hepatitis B.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20742
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; peginterferon alfa-2a

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]
- 2 (Experimental)
  Interventions: Drug: Entecavir; Drug: peginterferon alfa-2a [Pegasys]
- 3 (Experimental)
  Interventions: Drug: Entecavir; Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: Entecavir — 0.5mg po daily for 24 weeks
  Arms: 3
Drug: Entecavir — 0.5mg po daily from week 13 to week 36
  Arms: 2
Drug: peginterferon alfa-2a [Pegasys] — 180 micrograms sc/week for 48 weeks
  Arms: 1; 2
Drug: peginterferon alfa-2a [Pegasys] — 180 micrograms sc/week from week 21 to week 68
  Arms: 3

SUMMARY:
This 3 arm study will assess the efficacy and safety of PEGASYS + entecavir combination therapy in treatment-naive patients with HBeAg positive chronic hepatitis B. Patients will be randomized to receive 1)PEGASYS 180 micrograms s.c./week for 48 weeks, 2)PEGASYS 180 micrograms s.c./week for 48 weeks + entecavir 0.5mg p.o. once daily from week 13 to week 36 or 3) entecavir 0.5mg p.o. once daily for 24 weeks + PEGASYS 180 micrograms s.c./week from week 21 to 68. Treatment will be followed by 24 weeks treatment-free follow up. The anticipated time on study treatment is 3-12 months for groups 1 and 2, and 1-2 years for group 3, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-65 years of age;
* HBsAg positive, HBeAg positive and anti-HBe negative for at least 6 months, anti-HBs negative;
* absence of cirrhosis confirmed by liver biopsy in previous 12 months.

Exclusion Criteria:

* previous treatment for chronic hepatitis B within previous 6 months;
* antiviral, anti-neoplastic or immunomodulatory treatment in previous 6 months;
* co-infection with active hepatitis A, hepatitis C, hepatitis D or HIV;
* history or other evidence of a medical condition associated with chronic liver disease other than viral hepatitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2007-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Log change in quantitative HBeAg from baseline to 24 weeks after end of treatment. | Week 72 for Arms 1 and 2. Week 92 for Arm 3.

SECONDARY OUTCOMES:
HBeAg seroconversion, HBV-DNA <1000 copies/mL, loss of HBeAg, HBV DNA reduction, ALT normalization, loss of HBsAg seroconversion, reduction of HBsAg 24 weeks after end of treatment. | Week 72 for Arms 1 and 2. Week 92 for Arm 3.
AEs, laboratory parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- China (5):
  - Beijing
  - Hangzhou
  - Shanghai
  - Xi'an
  - Zhengzhou
- Hong Kong, Hong Kong

REFERENCES:
- [Derived] Xie Q, Zhou H, Bai X, Wu S, Chen JJ, Sheng J, Xie Y, Chen C, Chan HL, Zhao M. A randomized, open-label clinical study of combined pegylated interferon Alfa-2a (40KD) and entecavir treatment for hepatitis B "e" antigen-positive chronic hepatitis B. Clin Infect Dis. 2014 Dec 15;59(12):1714-23. doi: 10.1093/cid/ciu702. Epub 2014 Sep 4. PMID 25190434